CLINICAL TRIAL: NCT05185167
Title: Genotoxic Effects of Desflurane and Propofol Anesthesia in Patients Undergoing Lumbar Disc Surgery
Brief Title: Comparison of the Genotoxicity of Desflurane and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, Associate Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: MSKU 05/III
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: DNA Damage; Anesthesia
Keywords: Desflurane; Intravenous anesthetics; propofol; comet essay
MeSH Terms: interventions — Anesthetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desflurane Group (Experimental): Desflurane 1,0 minimum alveolar concentration will be administered during anesthesia maintenance
  Interventions: Drug: Anesthetics, General Desflurane Maintenance
- Propofol Group (Experimental): Propofol 6 mg//kg/hour will be administered during anesthesia maintenance
  Interventions: Drug: Anesthetics, General Propofol Maintenance

INTERVENTIONS:
Drug: Anesthetics, General Desflurane Maintenance — Comparison of dna damage of desflurane maintenance with propofol maintenance according to comet analysis
  Arms: Desflurane Group
Drug: Anesthetics, General Propofol Maintenance — Comparison of dna damage of propofol maintenance with desflurane maintenance according to comet analysis
  Arms: Propofol Group

SUMMARY:
The purpose of this study is to evaluate if the anesthetics propofol and desflurane can damage DNA according to comet essay in patients submitted to lumbar disc surgery.

DETAILED DESCRIPTION:
It is expected that DNA damage information provide the possible genotoxic effects of inhalational and intravenous anesthetics and contribute to the establishment of strategies aimed at reducing the risks to exposed patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent form
2. Elective lumbar spinal surgery that will take at least 120 minutes,
3. American Society of Anesthesiologists (ASA) physical status I and II

Exclusion Criteria:

1. Patients with ASA physical status III or IV disease
2. Chronic systemic disease (diabetes mellitus,chronic pulmonary disorders, chronic kidney and liver disorders)
3. Smoking or alcohol consumption
4. Recently received radiation, chemotherapy
5. Malignancy
6. Patients who will receive blood transfusion during the operation
7. Users of antioxidant supplements
8. Patients who have received general anesthesia in the last three months
9. Patients with known occupational exposures (operating room personnel, chemical plant worker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Intensity of the DNA tail detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | Before anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the intensity of the DNA tail, and the tail greater, the greater the damage.
Intensity of the DNA tail detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | 2 hours after anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the intensity of the DNA tail, and the tail greater, the greater the damage.
Intensity of the DNA tail detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 1st day
  The blood samples that evaluate with comet analysis aim to detect the intensity of the DNA tail, and the tail greater, the greater the damage.
Intensity of the DNA tail detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 5th day
  The blood samples that evaluate with comet analysis aim to detect the intensity of the DNA tail, and the tail greater, the greater the damage.
Head length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | Before anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the head length of DNA, the head greater, the smaller the damage.
Head length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | 2 hours after anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the head length of DNA, the head greater, the smaller the damage.
Head length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 1 st day
  The blood samples that evaluate with comet analysis aim to detect the head length of DNA, the head greater, the smaller the damage.
Head length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 5th day
  The blood samples that evaluate with comet analysis aim to detect the head length of DNA, the head greater, the smaller the damage.
Tail length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | before anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the tail length of DNA, the head greater, the greater the damage.
Tail length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | 2 hours after anesthesia induction
  The blood samples that evaluate with comet analysis aim to detect the tail length of DNA, the head greater, the greater the damage.
Tail length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 1 st day
  The blood samples that evaluate with comet analysis aim to detect the tail length of DNA, the head greater, the greater the damage.
Tail length of DNA detected by using Comet Assay IV Version 4.3.2 for Basler FireWire | postoperative 5th day
  The blood samples that evaluate with comet analysis aim to detect the tail length of DNA, the head greater, the greater the damage.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Korkmaz Toker, Assoc. Prof., Principal Investigator — Mugla Sıtkı Kocman University Department of Anesthesiology and reanimation
Locations (1):
- Mugla Sitki Kocman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toker MK, Altiparmak B, Gursoy G, Uysal AI, Dede G, Gundogdu G, Dodurga Y, Ugur B. Comparison of the genotoxicity of propofol and desflurane using the comet assay in the lymphocytes of patients who underwent lumbar discectomy: A randomized trial. Saudi Med J. 2024 May;45(5):468-475. doi: 10.15537/smj.2024.45.5.20240077. PMID 38734439